CLINICAL TRIAL: NCT00870870
Title: Randomized, Open Label, Stratified Phase 2 Trial of Gemcitabine, Carboplatin, and Cetuximab With Vs. Without IMC-A12 in Chemotherapy-Naive Patients With Advanced/Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of IMC-A12 (Cixutumumab) With and Without Other Standard Chemotherapies in Participants With Lung Cancer Who Have Not Received Chemotherapy Before
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13930; CP02-0860 (Other: CDER); CP13-0811 (Other: ImClone, LLC); I5A-IE-JAEF (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Results first posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Tumors; Antibodies, Monoclonal; Stage IIIb Metastatic Non-Small Cell Lung Cancer; Stage IV Metastatic Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Gemcitabine; Cisplatin; cixutumumab; Cetuximab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GCiC + IMC-A12 (Gemcitabine/Cisplatin/Cetuximab + Cixutumumab) (Experimental): Cycles repeat every 3 weeks for first 6 cycles (18 weeks) and then once every 2 weeks (maintenance therapy) until disease progression, intolerable toxicity, withdrawal of consent or other withdrawal criteria met
  *Cisplatin will replace Carboplatin. Gemcitabine/Carboplatin/Cetuximab (GCC) plus cixutumumab will change to Gemcitabine/Cisplatin/Cetuximab (GCiC) plus cixutumumab (participants enrolled subsequent to this change will receive gemcitabine, cisplatin and cetuximab, plus cixutumumab)
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Biological: IMC-A12 (cixutumumab); Biological: Cetuximab; Drug: Carboplatin
- GCiC (Gemcitabine/Cisplatin/Cetuximab) (Active Comparator): Cycles repeat every 3 weeks for 6 cycles (18 weeks) and then once every 2 weeks (maintenance therapy) until disease progression, intolerable toxicity, withdrawal of consent or other withdrawal criteria met
  *Cisplatin will replace Carboplatin. GCC plus cixutumumab will change to GCiC plus cixutumumab (participants enrolled subsequent to this change will receive gemcitabine, cisplatin and cetuximab, plus cixutumumab)
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Biological: Cetuximab; Drug: Carboplatin

INTERVENTIONS:
Drug: Gemcitabine — 1000 milligrams per square meter (mg/m^2) on Days 1 and 8 of each cycle
  [First 6 cycles (18 weeks)]
Drug: Cisplatin — 75 mg/m^2 on Day 1 of each cycle
  [First 6 cycles (18 weeks)]
Biological: IMC-A12 (cixutumumab) — 6 milligrams per kilogram (mg/kg) intravenous (IV) infusion, administered once per week (on Days 1, 8, and 15 of each cycle)
  [First 6 cycles (18 weeks)]
  Other Names: Cixutumumab; LY3012217
  Arms: GCiC + IMC-A12 (Gemcitabine/Cisplatin/Cetuximab + Cixutumumab)
Biological: Cetuximab — 400 mg/m^2 IV infusion, administered on Day 1 of Cycle 1, 250 mg/m^2 once per week thereafter
  [First 6 cycles (18 weeks)]
  Other Names: Erbitux®
Biological: IMC-A12 (cixutumumab) — 10 mg/kg IV infusion, administered once every 2 weeks
  (Maintenance therapy)
  Other Names: Cixutumumab; LY3012217
  Arms: GCiC + IMC-A12 (Gemcitabine/Cisplatin/Cetuximab + Cixutumumab)
Biological: Cetuximab — 500 mg/m^2 IV infusion, administered once every 2 weeks
  (Maintenance therapy)
  Other Names: Erbitux®
Drug: Carboplatin — Area under the curve (AUC) = 5, Day 1 of each cycle
  [First 6 cycles (18 weeks)]
  *Carboplatin will be replaced by Cisplatin

SUMMARY:
The purpose of this study is to determine the number of participants whose cancer shrinks or disappears after treatment on the study.

DETAILED DESCRIPTION:
Participants with Stage IIIb or IV non-small cell lung cancer (NSCLC) who have not received previous chemotherapy will be stratified, based on disease histology (squamous versus [vs.] nonsquamous).

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically confirmed, Stage IIIb - IV NSCLC
* Has metastatic disease
* Has a tumor measurable according to Response Evaluation Criteria in Solid Tumors (RECIST)
* Has adequate hematologic function
* Has adequate hepatic function
* Has adequate renal function
* Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation

Exclusion Criteria:

* Has uncontrolled brain metastases
* Has leptomeningeal disease
* Has received previous chemotherapy for NSCLC (participants who have received adjuvant chemotherapy are eligible if the last administration of the prior adjuvant regimen occurred at least 6 months prior to randomization)
* Receiving any other investigational agent(s)
* Has a history of treatment with other agents targeting the insulin-like growth factor (IGF) or the epidermal growth factor (EGF) receptor
* Has a known allergy / history of hypersensitivity reaction to any of the treatment components
* Has poorly controlled diabetes mellitus. Participants with a history of diabetes mellitus are allowed to participate, provided that their blood glucose is within normal range [fasting glucose <160 milligrams per deciliter (mg/dL) or below the upper limit of normal (ULN) and hemoglobin A1C≤ 7%] and that they are on a stable dietary or therapeutic regimen for this condition
* Has an uncontrolled intercurrent illness
* Pregnant or lactating
* Has a history of another primary cancer, with the exception of: a) curatively resected nonmelanomatous skin cancer; b) curatively treated cervical carcinoma in situ; or c) other primary solid tumor treated with curative intent and no known active disease present and no treatment administered during the last 3 years
* Has superior vena cava syndrome contraindicating hydration
* Has current clinically-relevant coronary artery disease (New York Heart Association III or IV) or uncontrolled congestive heart failure
* Has any National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE) Version (v) 3.0 Grade ≥2 peripheral neuropathy
* Has significant third space fluid retention, requiring repeated drainage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-03; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Director — Eli Lilly and Company
Locations (9):
- United States (9):
  - ImClone Investigational Site, Anniston, Alabama
  - ImClone Investigational Site, La Jolla, California
  - ImClone Investigational Site, Orange, California
  - ImClone Investigational Site, Orlando, Florida
  - ImClone Investigational Site, Atlanta, Georgia
  - ImClone Investigational Site, Chicago, Illinois
  - ImClone Investigational Site, Albuquerque, New Mexico
  - ImClone Investigational Site, New York, New York
  - ImClone Investigational Site, Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine/Carboplatin/Cetuximab (GCC): Gemcitabine: 1000 milligrams per square meter (mg/m^2) on Days 1 and 8 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Cetuximab: Initial dose of 400 mg/m^2 on Day 1 of Cycle 1, and subsequent doses of 250 mg/m^2 once every week (Q1W) of each 3-week cycle for a total of 6 cycles (18 weeks). Later administered at 500 mg/m^2 once every 2 weeks (Q2W) in the subsequent cycles (2-week cycles).
  Carboplatin: Area under the curve (AUC) = 5 on Day 1 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Treatment was continued until disease progression, unacceptable toxicity, withdrawal of consent or any other discontinuation criteria were met.
- GCC Plus Cixutumumab: Gemcitabine: 1000 mg/m^2 on Days 1 and 8 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Cetuximab: Initial dose of 400 mg/m^2 on Day 1 of Cycle 1 and subsequent doses of 250 mg/m^2 Q1W of each 3-week cycle for a total of 6 cycles (18 weeks). Later administered at 500 mg/m^2 Q2W in the subsequent cycles (2-week cycles).
  Carboplatin: AUC = 5 on Day 1 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Cixutumumab: 6 milligrams per kilogram (mg/kg) intravenous (IV) infusion Q1W on Days 1, 8, and 15 of each 3-week cycle for a total of 6 cycles (18 weeks). Later administered at 10 mg/kg IV Q2W in the subsequent cycles (2-week cycles).
  Treatment was continued until disease progression, unacceptable toxicity, withdrawal of consent or any other discontinuation criteria were met.
- Gemcitabine/Cisplatin/Cetuximab (GCiC): Gemcitabine: 1000 mg/m^2 on Days 1 and 8 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Cisplatin: 75 mg/m^2 on Day 1 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Cetuximab: Initial dose of 400 mg/m^2 on Day 1 of Cycle 1 and subsequent doses of 250 mg/m^2 Q1W of each 3-week cycle for a total of 6 cycles (18 weeks). Later administered at 500 mg/m^2 Q2W in the subsequent cycles (2-week cycles).
  Treatment was continued until disease progression, unacceptable toxicity, withdrawal of consent or any other discontinuation criteria were met.
- GCiC Plus Cixutumumab: Gemcitabine: 1000 mg/m^2 on Days 1 and 8 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Cisplatin: 75 mg/m^2 on Day 1 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Cetuximab: Initial dose of 400 mg/m^2 on Day 1 of Cycle 1 and subsequent doses of 250 mg/m^2 Q1W of each 3-week cycle for a total of 6 cycles (18 weeks). Later administered at 500 mg/m^2 Q2W in the subsequent cycles (2-week cycles).
  Cixutumumab: 6 mg/kg IV infusion Q1W on Days 1, 8, and 15 of each 3-week cycle for a total of 6 cycles (18 weeks). Later administered at 10 mg/kg IV Q2W in the subsequent cycles (2-week cycles).
  Treatment was continued until disease progression, unacceptable toxicity, withdrawal of consent or any other discontinuation criteria were met.
Period: Overall Study
Arm/Group | Gemcitabine/Carboplatin/Cetuximab (GCC) | GCC Plus Cixutumumab | Gemcitabine/Cisplatin/Cetuximab (GCiC) | GCiC Plus Cixutumumab
Started | 4 | 6 | 29 | 25
Completed | 4 | 5 | 26 | 20
Not Completed | 0 | 1 | 3 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Gemcitabine/Carboplatin/Cetuximab (GCC): Gemcitabine: 1000 mg/m^2 on Days 1 and 8 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Cetuximab: Initial dose of 400 mg/m^2 on Day 1 of Cycle 1, and subsequent doses of 250 mg/m^2 Q1W of each 3-week cycle for a total of 6 cycles (18 weeks). Later administered at 500 mg/m^2 Q2W in the subsequent cycles (2-week cycles).
  Carboplatin: AUC = 5 on Day 1 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Treatment was continued until disease progression, unacceptable toxicity, withdrawal of consent or any other discontinuation criteria were met.
- GCC Plus Cixutumumab: Gemcitabine: 1000 mg/m^2 on Days 1 and 8 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Cetuximab: Initial dose of 400 mg/m^2 on Day 1 of Cycle 1, and subsequent doses of 250 mg/m^2 Q1W of each 3-week cycle for a total of 6 cycles (18 weeks). Later administered at 500 mg/m^2 Q2W in the subsequent cycles (2-week cycles).
  Carboplatin: AUC = 5 on Day 1 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Cixutumumab: 6 mg/kg IV infusion Q1W on Days 1, 8, and 15 of each 3-week cycle for a total of 6 cycles (18 weeks). Later administered at 10 mg/kg IV Q2W in the subsequent cycles (2-week cycles).
  Treatment was continued until disease progression, unacceptable toxicity, withdrawal of consent or any other discontinuation criteria were met.
- Gemcitabine/Cisplatin/Cetuximab (GCiC): Gemcitabine: 1000 mg/m^2 on Days 1 and 8 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Cisplatin: 75 mg/m^2 on Day 1 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Cetuximab: Initial dose of 400 mg/m^2 on Day 1 of Cycle 1, and subsequent doses of 250 mg/m^2 Q1W of each 3-week cycle for a total of 6 cycles (18 weeks). Later administered at 500 mg/m^2 Q2W in the subsequent cycles (2-week cycles).
  Treatment was continued until disease progression, unacceptable toxicity, withdrawal of consent or any other discontinuation criteria were met.
- GCiC Plus Cixutumumab: Gemcitabine: 1000 mg/m^2 on Days 1 and 8 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Cisplatin: 75 mg/m^2 on Day 1 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Cetuximab: Initial dose of 400 mg/m^2 on Day 1 of Cycle 1, and subsequent doses of 250 mg/m^2 Q1W of each 3-week cycle for a total of 6 cycles (18 weeks). Later administered at 500 mg/m^2 Q2W in the subsequent cycles (2-week cycle).
  Cixutumumab: 6 mg/kg IV infusion Q1W on Days 1, 8, and 15 of each 3-week cycle for a total of 6 cycles (18 weeks). Later administered at 10 mg/kg IV Q2W in the subsequent cycles (2-week cycles).
  Treatment was continued until disease progression, unacceptable toxicity, withdrawal of consent or any other discontinuation criteria were met.
- Total: Total of all reporting groups
Arm/Group | Gemcitabine/Carboplatin/Cetuximab (GCC) | GCC Plus Cixutumumab | Gemcitabine/Cisplatin/Cetuximab (GCiC) | GCiC Plus Cixutumumab | Total
Number analyzed (Participants) | 4 | 6 | 29 | 25 | 64
Age, Continuous [Median (Full Range); unit: years] | 68.50 [65.00 to 74.00] | 54.50 [49.00 to 69.00] | 64.00 [45.00 to 77.00] | 60.00 [41.00 to 77.00] | 62.00 [41.00 to 77.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 13 | 11 | 27
  Male | 3 | 4 | 16 | 14 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 6 | 29 | 24 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 6 | 26 | 22 | 58
  Black or African American | 0 | 0 | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 6 | 29 | 25 | 64
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 173.10 (3.982) | 176.78 (8.935) | 170.04 (9.356) | 167.79 (10.537) | 169.99 (9.758)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 74.93 (13.814) | 80.43 (16.720) | 76.30 (13.908) | 72.90 (15.957) | 75.27 (14.815)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: square meters (m^2)] — BSA is the measured or calculated surface area of a human body based on body weight and height.
  square meters (m^2) | 1.89 (0.186) | 1.98 (0.223) | 1.89 (0.214) | 1.84 (0.246) | 1.88 (0.225)
Eastern Cooperative Oncology Status Performance Status (ECOG PS) Score [Count of Participants; unit: Participants] — ECOG performance status was used to classify participants according to their functional impairment. Score 0 = fully active, able to carry on all pre-disease performance without restriction. Score 1 = restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, for example, light house work, office work.
  Participants
    0 = Fully Active | 0 | 4 | 5 | 9 | 18
    1 = Ambulatory, Restricted Work Activity | 4 | 2 | 24 | 16 | 46
Randomization Stratum [Count of Participants; unit: Participants]
  Squamous | 2 | 3 | 14 | 11 | 30
  Nonsquamous | 2 | 3 | 15 | 14 | 34

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) [Objective Response Rate (ORR)]
Description: ORR was defined as the percentage of participants achieving either CR or PR. Response was defined using Response Evaluation Criteria in Solid Tumors (RECIST), version (v) 1.0 criteria. CR was defined as the disappearance of all target and non-target lesions and the normalization of the tumour marker level. PR was defined as having at least a 30% decrease in sum of longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Percentage of participants is calculated as a total number of participants with CR or PR / total number of participants treated * 100.
Time Frame: Randomization to measured progressive disease (PD) (up to 16.9 months)
Population: All participants randomized to GCiC and GCiC Plus Cixutumumab arms. Efficacy data were not summarized for the original treatment arms (GCC and GCC Plus Cixutumumab) since such summaries were not considered relevant to the study objectives under the amended protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- GCiC Plus Cixutumumab: Gemcitabine: 1000 mg/m^2 on Days 1 and 8 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Cisplatin: 75 mg/m^2 on Day 1 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Cetuximab: Initial dose of 400 mg/m^2 on Day 1 of Cycle 1, and subsequent doses of 250 mg/m^2 Q1W of each 3-week cycle for a total of 6 cycles (18 weeks). Later administered at 500 mg/m^2 Q2W in the subsequent cycles (2-week cycles).
  Cixutumumab: 6 mg/kg IV infusion Q1W on Days 1, 8, and 15 of each 3-week cycle for a total of 6 cycles (18 weeks). Later administered at 10 mg/kg IV Q2W in the subsequent cycles (2-week cycles).
  Treatment was continued until disease progression, unacceptable toxicity, withdrawal of consent or any other discontinuation criteria were met.
Arm/Group | Gemcitabine/Cisplatin/Cetuximab (GCiC) | GCiC Plus Cixutumumab
Number analyzed (Participants) | 29 | 25
percentage of participants | 31.0 [14.2 to 47.9] | 20.0 [4.3 to 35.7]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the duration from the date of randomization to the date of death from any cause. For participants who were alive, OS was censored at the date of last follow-up visit or at the date of last contact.
Time Frame: Randomization to death due to any cause or censor (up to 30.4 months)
Population: All participants randomized to GCiC and GCiC Plus Cixutumumab arms. Participants censored: GCiC = 6, GCiC Plus cixutumumab = 6. Efficacy data were not summarized for the original treatment arms (GCC and GCC Plus Cixutumumab) since such summaries were not considered relevant to the study objectives under the amended protocol.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- GCiC: Gemcitabine: 1000 mg/m^2 on Days 1 and 8 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Cisplatin: 75 mg/m^2 on Day 1 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Cetuximab: Initial dose of 400 mg/m^2 on Day 1 of Cycle 1, and subsequent doses of 250 mg/m^2 Q1W of each 3-week cycle for a total of 6 cycles (18 weeks). Later administered at 500 mg/m^2 Q2W in the subsequent cycles (2-week cycles).
  Treatment was continued until disease progression, unacceptable toxicity, withdrawal of consent or any other discontinuation criteria were met.
Arm/Group | GCiC | GCiC Plus Cixutumumab
Number analyzed (Participants) | 29 | 25
months | 11.5 [5.3 to 14.8] | 8.9 [7.0 to 13.2]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the duration from the date of randomization until disease progression or death due to any cause, whichever occurred first. Response was defined using RECIST, v 1.0 criteria. PD was defined as having a ≥20% increase in sum of LD of target lesions or the appearance of new lesions and/or unequivocal progression of non-target lesions. For participants who were alive and without disease progression, PFS was censored at the date of last objective tumor assessment. For participants who did not experience disease progression and were lost to follow-up, PFS was censored at the date of the last objective tumor assessment or the date of last contact.
Time Frame: Randomization to PD or death due to any cause or censor (up to 16.9 months)
Population: All participants randomized to GCiC and GCiC Plus Cixutumumab arms. Participants censored: GCiC = 2, GCiC Plus cixutumumab = 10. Efficacy data were not summarized for the original treatment arms (GCC and GCC Plus Cixutumumab) since such summaries were not considered relevant to the study objectives under the amended protocol.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GCiC | GCiC Plus Cixutumumab
Number analyzed (Participants) | 29 | 25
months | 4.2 [2.9 to 6.2] | 5.6 [2.6 to 7.0]

4. Secondary Outcome: Time To Progression (TTP)
Description: TTP was defined as the duration from the date of randomization until the date of disease progression. Response was defined using RECIST v 1.0 criteria. PD was defined as having a ≥20% increase in the sum of LD of target lesions or the appearance of new lesions and/or unequivocal progression of non-target lesions. For participants without disease progression, TTP was censored at the date of last objective tumor assessment. For participants without disease progression and were subsequently lost to follow-up, TTP was censored at the date of last follow-up visit or at the date of last contact.
Time Frame: Randomization to months until PD or censor (up to 16.9 months)
Population: All participants (pts) randomized to GCiC and GCiC Plus Cixutumumab arms. Participants censored: GCiC = 9, GCiC Plus Cixutumumab = 12. Efficacy data were not summarized for the original treatment arms (GCC and GCC Plus Cixutumumab) since such summaries were not considered relevant to the study objectives under the amended protocol.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GCiC | GCiC Plus Cixutumumab
Number analyzed (Participants) | 29 | 25
months | 5.8 [3.9 to 6.7] | 5.7 [2.7 to 11.7]

5. Secondary Outcome: Duration of Response
Description: The duration of CR or PR was defined as the time from first objective status assessment of CR or PR to the first time of disease progression or death. Response was defined using RECIST v 1.0 criteria. CR was defined as the disappearance of all target lesions and non-target lesions. PR was defined as having at least a 30% decrease in sum of LD of target lesions. Duration of response was censored on the date of last tumor assessment for participants who were alive and have no evidence of disease progression.
Time Frame: Date of first response to the date of PD or death due to any cause or censor ( up to 15.5 months)
Population: All pts randomized to GCiC and GCiC Plus Cixutumumab arms and who had CR or PR, except 1 pt in GCiC group eliminated d/t PR after starting additional treatment. Participants censored: GCiC = 0, GCiC Plus Cixutumumab = 1. Efficacy data were not summarized for the original treatment arms (GCC and GCC Plus Cixutumumab) due to the amended protocol.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GCiC | GCiC Plus Cixutumumab
Number analyzed (Participants) | 8 | 4
months | 4.8 [4.2 to 5.3] | 4.8 [2.9 to 15.5]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs) or Deaths
Description: Data presented are the number of participants who experienced 1 or more AEs, serious AEs (SAEs), and AEs that lead to death during the study including the 30-day follow-up. A summary of SAEs and other non-serious AEs, regardless of causality is located in the Reported Adverse Events section of this report.
Time Frame: Randomization to last dose of study medication (up to 11.7 months) plus 30-day safety follow-up
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine/Carboplatin/Cetuximab (GCC) | GCC Plus Cixutumumab | Gemcitabine/Cisplatin/Cetuximab (GCiC) | GCiC Plus Cixutumumab
Number analyzed (Participants) | 4 | 6 | 29 | 25
Participants
  AEs | 4 | 6 | 29 | 25
  SAEs | 4 | 5 | 20 | 15
  Deaths Due to AEs | 1 | 1 | 4 | 1

7. Secondary Outcome: Serum Anti-Cixutumumab Antibody Assessment (Immunogenicity)
Time Frame: Prior to first infusions of Cycles 1, 3, and 5 and 30 days following the end of therapy
Population: Zero participants analyzed. Analysis was not performed due to lack of an appropriate validated assay.
Arm/Group | GCC Plus Cixutumumab | GCiC Plus Cixutumumab
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Maximum Concentration (Cmax) of Cixutumumab at Study Day 1
Time Frame: Day 1
Population: Zero participants analyzed. No PK samples analyzed due to being expired prior to assay developed to analyze.
Arm/Group | GCC Plus Cixutumumab | GCiC Plus Cixutumumab
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Cmax of Cixutumumab for Cycle 1
Time Frame: Week 1 (Cycle 1, Day 1)
Population: Zero participants analyzed. No PK samples analyzed due to being expired prior to assay developed to analyze.
Arm/Group | GCC Plus Cixutumumab | GCiC Plus Cixutumumab
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Cmax of Cixutumumab for Cycle 3
Time Frame: Week 7 (Cycle 3, Day 1)
Population: Zero participants analyzed. No PK samples analyzed due to being expired prior to assay developed to analyze.
Arm/Group | GCC Plus Cixutumumab | GCiC Plus Cixutumumab
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Cmax of Cixutumumab Cycle 5
Time Frame: Week 13 (Cycle 5, Day 1)
Population: Zero participants analyzed. No PK samples analyzed due to being expired prior to assay developed to analyze.
Arm/Group | GCC Plus Cixutumumab | GCiC Plus Cixutumumab
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Minimum Concentration (Cmin) of Cixutumumab at Study Day 1
Time Frame: Day 1
Population: Zero participants analyzed. No PK samples analyzed due to being expired prior to assay developed to analyze.
Arm/Group | GCC Plus Cixutumumab | GCiC Plus Cixutumumab
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Cmin of Cixutumumab for Cycle 1
Time Frame: Week 1 (Cycle 1, Day 1)
Population: Zero participants analyzed. No PK samples analyzed due to being expired prior to assay developed to analyze.
Arm/Group | GCC Plus Cixutumumab | GCiC Plus Cixutumumab
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Cmin of Cixutumumab for Cycle 3
Time Frame: Week 7 (Cycle 3, Day 1)
Population: Zero participants analyzed. No PK samples analyzed due to being expired prior to assay developed to analyze.
Arm/Group | GCC Plus Cixutumumab | GCiC Plus Cixutumumab
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Cmin of Cixutumumab for Cycle 5
Time Frame: Week 13 (Cycle 5, Day 1)
Population: Zero participants analyzed. No PK samples analyzed due to being expired prior to assay developed to analyze.
Groups:
- GCiC Plus Cixutumumab: Gemcitabine: 1000 mg/m^2 on Days 1 and 8 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Cisplatin: 75 mg/m^2 on Day 1 of each 3-week cycle for a total of 6 cycles (18 weeks).
  Cetuximab: Initial dose of 400 mg/m^2 on Day 1 of Cycle 1, and subsequent doses of 250 mg/m^2 Q1W of each 3-week cycle for a total of 6 cycles (18 weeks). Later administered at 500 mg/m^2 Q2W in the subsequent cycles (2-week cycle).
  Cixutumumab: 6 mg/kg IV infusion Q1W on Days 1, 8, and 15 of each 3-week cycle for a total of 6 cycles (18 weeks). Later administered at 10 mg/kg Q2W in the subsequent cycles (2-week cycle).
  Treatment was continued until disease progression, unacceptable toxicity, withdrawal of consent or any other discontinuation criteria were met.
Arm/Group | GCC Plus Cixutumumab | GCiC Plus Cixutumumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Gemcitabine/Carboplatin/Cetuximab (GCC) | GCC Plus Cixutumumab | Gemcitabine/Cisplatin/Cetuximab (GCiC) | GCiC Plus Cixutumumab
Serious Adverse Events (participants affected / at risk) | 4/4 | 5/6 | 20/29 | 15/25
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6 | 29/29 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine/Carboplatin/Cetuximab (GCC) (N=4) | GCC Plus Cixutumumab (N=6) | Gemcitabine/Cisplatin/Cetuximab (GCiC) (N=29) | GCiC Plus Cixutumumab (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (6) | 4 (5) | 2 (2) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gallbladder non-functioning (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection pseudomonas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (4) | 3 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Gemcitabine/Carboplatin/Cetuximab (GCC) (N=4) | GCC Plus Cixutumumab (N=6) | Gemcitabine/Cisplatin/Cetuximab (GCiC) (N=29) | GCiC Plus Cixutumumab (N=25)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 10 (31) | 9 (27)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (3) | 4 (7) | 17 (44) | 12 (22)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (4) | 2 (5) | 18 (42) | 19 (55)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 5 (9) | 2 (2)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 4 (7)
Constipation (Gastrointestinal disorders) | 2 (6) | 2 (6) | 17 (25) | 17 (26)
Diarrhoea (Gastrointestinal disorders) | 4 (7) | 2 (5) | 13 (20) | 9 (22)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (11) | 3 (5) | 15 (35) | 15 (28)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 3 (8) | 11 (18) | 15 (21)
Vomiting (Gastrointestinal disorders) | 2 (4) | 0 (0) | 9 (13) | 6 (8)
Asthenia (General disorders) | 0 (0) | 0 (0) | 3 (4) | 3 (4)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Catheter thrombosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Early satiety (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (18) | 4 (12) | 21 (28) | 17 (34)
Infusion related reaction (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 5 (9) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Incision site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 3 (5) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 1 (2) | 2 (8) | 5 (9)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Blood amylase increased (Investigations) | 1 (2) | 0 (0) | 2 (3) | 2 (3)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 3 (4) | 4 (5)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 4 (16) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 3 (4) | 2 (6)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 12 (15) | 9 (10)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 2 (5) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 10 (16) | 10 (14)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 6 (11) | 7 (21)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (5) | 1 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 6 (14) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 7 (11) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 14 (49) | 9 (22)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (7) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (4) | 3 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 5 (7) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 5 (5) | 3 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (2) | 5 (6) | 4 (4)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 8 (14) | 4 (5)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 8 (9) | 6 (7)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (2) | 7 (11) | 4 (6)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Prostatitis (Reproductive system and breast disorders) | 0/3 (0) | 1/4 (1) | 0/16 (0) | 0/14 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 3 (6) | 5 (6) | 5 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (7) | 7 (9) | 4 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (5) | 9 (12) | 15 (20)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 6 (6) | 7 (8)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 (8) | 5 (12) | 12 (21) | 8 (12)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 5 (7) | 9 (13)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 14 (25) | 17 (35)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 7 (12) | 12 (14)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 6 (6) | 2 (2)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.